CLINICAL TRIAL: NCT01824875
Title: A Randomized Phase II Study of Temozolomide or Temozolomide and Capecitabine in Patients With Advanced Pancreatic Neuroendocrine Tumors
Brief Title: Temozolomide With or Without Capecitabine in Treating Patients With Advanced Pancreatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2211; NCI-2012-02007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E2211 (Other: ECOG-ACRIN Cancer Research Group); U10CA021115 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Islet Cell Carcinoma; Pancreatic Polypeptide Tumor; Recurrent Islet Cell Carcinoma; Somatostatinoma
Keywords: temozolomide; capecitabine; pancreatic neuroendocrine tumor
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Somatostatinoma; Adenoma, Islet Cell | interventions — Temozolomide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide
- Arm B (temozolomide and capecitabine) (Experimental): Patients receive capecitabine PO BID on days 1-14 and temozolomide PO QD on days 10-14. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide; Drug: capecitabine

INTERVENTIONS:
Drug: temozolomide — Given PO
  Other Names: Temodar
Drug: capecitabine — Given PO
  Other Names: Xeloda
  Arms: Arm B (temozolomide and capecitabine)

SUMMARY:
This randomized phase II trial studies how well giving temozolomide with or without capecitabine works in treating patients with advanced pancreatic neuroendocrine tumors. Drugs used in chemotherapy, such as temozolomide and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether temozolomide is more effective with or without capecitabine in treating patients with advanced pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) associated with temozolomide alone or temozolomide and capecitabine in patients with advanced pancreatic neuroendocrine tumors.

SECONDARY OBJECTIVES:

I. To evaluate response rates (RR) associated with temozolomide alone or temozolomide and capecitabine treatment in patients with advanced pancreatic neuroendocrine tumors.

II. To evaluate overall survival (OS) associated with temozolomide alone or temozolomide and capecitabine in patients with advanced pancreatic neuroendocrine tumors.

III. To evaluate the toxicity associated with temozolomide alone or temozolomide and capecitabine treatment in patients with advanced pancreatic neuroendocrine tumors.

IV. To evaluate the usefulness of methyl guanine methyltransferase (MGMT) status (by immunohistochemistry [IHC] and promoter methylation) for predicting response in pancreatic neuroendocrine tumor patients treated with either temozolomide or temozolomide and capecitabine.

V. To bank radiology images for evaluation of quality, reproducibility, and compliance with computed tomography (CT) methodology.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive temozolomide orally (PO) once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive capecitabine PO twice daily (BID) on days 1-14 and temozolomide PO QD on days 10-14. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or pathologically confirmed locally unresectable or metastatic low or intermediate grade pancreatic neuroendocrine tumor
* Patient must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria; baseline measurements and evaluations of all sites of disease must be obtained <= 4 weeks prior to randomization and must be acquired by multiphasic CT or contrast magnetic resonance imaging (MRI)
* Date of last documented disease progression must be within 12 months from date of randomization
* Prior everolimus and/or sunitinib therapy is allowed, so long as it was discontinued >= 4 weeks prior to randomization
* Concurrent somatostatin analogues are allowed provided that patients

  * Have been on a stable dose for 8 weeks and
  * Have documented disease progression on that dose
* Chemoembolization is allowed if ≥ 4 weeks from study entry. There are 2 possible scenarios:

  * If patient has hepatic disease only: they need to have progressed in the liver since chemoembolization and have measurable disease by RECIST 1.1 in order to be eligible.
  * If patient has hepatic and extrahepatic disease: they will need to have progressed inside OR outside the liver and have measureable disease by RECIST 1.1 in order to be eligible.
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mm^3
* Total bilirubin <= institutional upper limit of normal (ULN) or <= 1.5 X institutional ULN (if the patient has liver metastases)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) <= 3 X institutional ULN or (<= 5 X institutional ULN if the patient has liver metastases)
* Serum creatinine <= 1.5 X institutional ULN
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must have life expectancy >= 12 weeks all females of childbearing potential must have a blood test or urine study within =< 2 weeks prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study; should a woman become pregnant while participating in this study, she should inform her treating physician immediately; if a man impregnates a woman while participating in this study, he should inform his treating physician immediately
* Patient must be able to swallow pills
* Patient must be able to tolerate CT or magnetic resonance (MR) imaging including contrast agents as required for their treatment and the protocol

Exclusion Criteria:

* Small cell carcinoma
* Prior temozolomide, dacarbazine (DTIC), or capecitabine, or 5-FU (fluorouracil) therapy
* Receiving any other investigational agents while on study treatment
* Receiving Coumadin while on treatment; other anticoagulants are allowed
* Patients with either clinically apparent central nervous system metastases or carcinomatous meningitis are ineligible
* Active or uncontrolled infection or serious medical or psychiatric illness
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or capecitabine
* Absorption issues that would limit the ability to absorb study agents
* Patients with a history of the following within 12 months of study entry:

  * Arterial thromboembolic events
  * Unstable angina
  * Myocardial Infarction
* Symptomatic peripheral vascular disease
* Patients with previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, or breast cancer in situ OR
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years OR
  * Prior malignancy cured by non-surgical modalities and patient has been continuously disease free for > 5 years
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-08-08 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Kunz, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (323):
- United States (323):
  - Kaiser Anaheim Medical Center, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Medical Group - Baldwin Park, Baldwin Park, California
  - Kaiser Foundation Hospital, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Southern California Permanente Medical Group, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Kaiser Permanente-West Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente Medical Center, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente at San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF-Mount Zion, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente Health Care, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Edna Williams Cancer Center at the Baptist Cancer Institute, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Galesburg Cottage Plaza Office, Galesburg, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Incorporated, Crestview Hills, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - New York Oncology Hematology PC - Amsterdam, Amsterdam, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - New York Oncology Hematology PC - Latham, Latham, New York
  - New York Oncology Hematology PC - Rexford, Rexford, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Weiler Division, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology and Hematology Care Incorporated, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Oncology and Hematology Care Inc - Blue Ash, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Western Hills, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center-Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute/Greenville CCOP, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Kunz PL, Graham NT, Catalano PJ, Nimeiri HS, Fisher GA, Longacre TA, Suarez CJ, Martin BA, Yao JC, Kulke MH, Hendifar AE, Shanks JC, Shah MH, Zalupski MM, Schmulbach EL, Reidy-Lagunes DL, Strosberg JR, O'Dwyer PJ, Benson AB 3rd. Randomized Study of Temozolomide or Temozolomide and Capecitabine in Patients With Advanced Pancreatic Neuroendocrine Tumors (ECOG-ACRIN E2211). J Clin Oncol. 2023 Mar 1;41(7):1359-1369. doi: 10.1200/JCO.22.01013. Epub 2022 Oct 19. PMID 36260828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on April 11, 2013 and closed on March 7, 2016 for a total of 144 patients enrolled. The first patient was accrued on August 8, 2013.
Period: Overall Study
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine)
Started | 72 | 72
Received Treatment and Adverse Event Data Available | 68 | 71
Eligible | 65 | 68
Eligible Patients With MGMT by IHC Data Available | 47 | 50
Eligible Patients With MGMT by Promoter Methylation Data Available | 27 | 30
Completed | 26 | 32
Not Completed | 46 | 40
Not completed — Disease progression | 22 | 15
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Adverse Event | 4 | 10
Not completed — Alternative therapy | 3 | 0
Not completed — Complicating disease | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Non-compliance | 1 | 1
Not completed — Treatment ended early due to mis-interpretation of protocol | 1 | 0
Not completed — Administrative issues | 0 | 2
Not completed — Ineligible or never started treatment | 9 | 5
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Only eligible patients were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine) | Total
Number analyzed (Participants) | 65 | 68 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.5) | 61.0 (10.9) | 60.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 35 | 38 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 60 | 63 | 123
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 5 | 17
  White | 50 | 56 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is defined as the time from randomization to progression or death without evidence of progression. Progression was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Kaplan-Meier method was used to estimate PFS.
Time Frame: Assessed every 3 months for 3 years and then every 6 months for years 3-5
Population: Only eligible patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine)
Number analyzed (Participants) | 65 | 68
months | 15.1 [10.5 to 21.0] | 23.2 [16.6 to 32.2]
Statistical Analysis 1: Comparison: Arm A (Temozolomide) vs Arm B (Temozolomide and Capecitabine); Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.46 to 1.07] — Hazard ratio of Arm B/Arm A

2. Secondary Outcome: Proportion of Patients With Response
Description: Response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and defined as either complete response (CR) or partial response (PR).
  CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed every 3 months for 3 years and then every 6 months for years 3-5
Population: Only eligible patients were included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine)
Number analyzed (Participants) | 65 | 68
proportion of participants | 0.338 [0.241 to 0.447] | 0.397 [0.297 to 0.504]
Statistical Analysis 1: Comparison: Arm A (Temozolomide) vs Arm B (Temozolomide and Capecitabine); Test type: Superiority; p = 0.59, Fisher Exact

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 3 years and then every 6 months for years 3-5
Population: Only eligible patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine)
Number analyzed (Participants) | 65 | 68
months | 53.8 [35.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 58.7 [44.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Association Between Methyl Guanine Methyltransferase (MGMT) Status by Immunohistochemistry (IHC) and Response
Description: Response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and defined as either complete response (CR) or partial response (PR). CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  MGMT status was determined by IHC using paraffin-embedded sections of 4µm. A score (H-score) was generated based on the findings and scoring was performed by two pathologists. This H-score ranges from 0 (no staining in the tumor) to 300 (diffuse intense staining of the tumor). The highest score was used if there was disagreement. H-scores were grouped into 3 standard categories for MGMT status:
  Category 1 - <=50 Category 2 - 51-100 Category 3 - >100
Time Frame: Assessed every 3 months for 3 years and then every 6 months for years 3-5
Population: Only eligible patients with MGMT status by IHC data available were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- MGMT by IHC: 1-2: MGMT status was determined by IHC and was categorized as IHC of 1-2.
- MGMT by IHC: 3: MGMT status was determined by IHC and was categorized as IHC of 3.
Arm/Group | MGMT by IHC: 1-2 | MGMT by IHC: 3
Number analyzed (Participants) | 63 | 34
Participants
  No response | 30 | 29
  Response | 33 | 5

5. Secondary Outcome: Association Between Methyl Guanine Methyltransferase (MGMT) Status by Promoter Methylation and Response
Description: Response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) and defined as either complete response (CR) or partial response (PR).
  CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  MGMT status is determined by promoter methylation, a clinically validated methylation-specific polymerase chain reaction (PCR) analysis. A tumor sample is considered positive for MGMT promoter methylation if an 80bp band is detected in the methylated PCR reaction. It would be considered MGMT negative if an 80bp band is not detected in the methylated PCR reaction.
Time Frame: Assessed every 3 months for 3 years and then every 6 months for years 3-5
Population: Only eligible patients with MGMT by promoter methylation data available were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- MGMT Negative: MGMT status was determined by promoter methylation and was categorized as negative.
- MGMT Positive: MGMT status was determined by promoter methylation and was categorized as positive.
Arm/Group | MGMT Negative | MGMT Positive
Number analyzed (Participants) | 50 | 7
Participants
  No response | 31 | 1
  Response | 19 | 6

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Description: All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
Groups:
- Arm A (Temozolomide): ARM A: Patients receive temozolomide orally (PO) once daily (QD) on days 1-5. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Temozolomide and Capecitabine): ARM B: Patients receive capecitabine PO twice daily (BID) on days 1-14 and temozolomide PO QD on days 10-14. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Temozolomide) | Arm B (Temozolomide and Capecitabine)
All-Cause Mortality (participants affected / at risk) | 42/72 | 33/72
Serious Adverse Events (participants affected / at risk) | 15/68 | 32/71
Other Adverse Events (participants affected / at risk) | 63/68 | 70/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Temozolomide) (N=68) | Arm B (Temozolomide and Capecitabine) (N=71)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Fatigue (General disorders) | 1 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 6
Lung infection (Infections and infestations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 5
Neutrophil count decreased (Investigations) | 3 | 9
Platelet count decreased (Investigations) | 7 | 7
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Temozolomide) (N=68) | Arm B (Temozolomide and Capecitabine) (N=71)
Anemia (Blood and lymphatic system disorders) | 21 | 27
Fatigue (General disorders) | 44 | 45
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 23
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 12
Abdominal pain (Gastrointestinal disorders) | 12 | 13
Constipation (Gastrointestinal disorders) | 22 | 34
Diarrhea (Gastrointestinal disorders) | 16 | 30
Mucositis oral (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 41 | 51
Vomiting (Gastrointestinal disorders) | 20 | 28
Skin infection (Infections and infestations) | 0 | 4
Blood bilirubin increased (Investigations) | 1 | 10
Lymphocyte count decreased (Investigations) | 0 | 5
Neutrophil count decreased (Investigations) | 7 | 13
Platelet count decreased (Investigations) | 25 | 24
Anorexia (Metabolism and nutrition disorders) | 14 | 13
Headache (Nervous system disorders) | 18 | 10
Lethargy (Nervous system disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/75/NCT01824875/Prot_SAP_000.pdf